CLINICAL TRIAL: NCT06750055
Title: Comparison of Walking With Wearable Gait Analysis System in Patients Undergoing Lumbar Spinal Stenosis Surgery
Brief Title: Gait Assessment in Lumbar Spinal Stenosis
Status: Recruiting | Type: Observational
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Fatma OZ, research assistant, Pamukkale University
Other Study IDs: FOZ
Record Dates: First submitted 2024-12-19; First posted 2024-12-27 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Lumbar Spinal Stenosis
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- lumbar spinal stenosis patient group: Assessment of Disability Status (Oswestry Disability Index) Pain Assessment (Visual Analog Scale-VAS) Quality of Life Assessment (SF-12) Evaluation of Gait Parameters: 10 Meter Walk Test-BTS G-Walk gait analysis system
- healthy control group: Quality of Life Assessment (SF-12) Evaluation of Gait Parameters: 10 Meter Walk Test-BTS G-Walk gait analysis system

SUMMARY:
Lumbar spinal stenosis (LSS) is a clinical condition in which the structures within the canal are compressed as a result of the narrowing of the lumbar spinal canal and nerve root canals, which is often caused by bones and soft tissues, causing back pain and neurological deficits in the lower extremities. The incidence in the general population has been reported as 1.7-8%. It begins to be seen after the age of 50 and its incidence increases after the age of 65. According to studies, LSS has been detected in 5% of patients who apply to a general practitioner with persistent back pain. Although it can be congenital, most cases of lumbar spinal stenosis are caused by changes in the aging spine as a result of degenerative processes. Changes that can lead to lumbar spinal stenosis include facet joint hypertrophy, decreased intervertebral disc height, osteophyte formation and ligamentum flavum hypertrophy. Clinical findings of LSS include symptoms such as back pain, leg pain, paresthesia, weakness and neurogenic claudication. Patients with neurogenic claudication experience increased pain when walking and standing and decreased pain when bending forward. Patients with LSS often change their spinal posture to allow more lumbar flexion to minimize pain and symptoms while walking; this can lead to gait abnormalities.

Walking function is important for the maintenance of daily living activities. Gait disturbance is associated with poor health outcomes. In a gait cycle, the foot has two distinct phases: stance and swing. These gait phases can be analyzed as a proportion of the gait cycle and compared to normative values. Furthermore, with the use of more advanced systems and devices, it is also possible to assess asymmetries and gait variability in the pelvis and other structures during gait.

Technological advances have led to the emergence of reliable surface sensor technologies capable of gait analysis in the form of wearable accelerometers. These devices provide continuous and objective data streams, including parameters such as daily step count, step rate, and step length. Numerous studies have investigated walking function in LSS patients using various devices including motion capture systems, inertial sensors, accelerometers, wearable technologies, electromyography (EMG) and force platforms. In the study, walking impairment in LSS patients compared to healthy participants was a significant decrease in walking speed and step length, a slight decrease in cadence and a slight increase in step duration. As the double-step support and stance phase ratios increase, the swing phase ratio decreases. Walking asymmetry between the feet also increases in all phases including stance, swing and double-step support. In addition, LSS patients may exhibit gait variability with each step. The reasons for these changing gait patterns are thought to be radicular pain, muscle weakness, low walking tolerance and increased instability with lumbar spine posture in the lumbar extension position during walking.

Winter et al. evaluated the walking ability in daily life in patients with knee or hip osteoarthritis and lumbar spinal stenosis with the help of a wearable accelerometer device. As a result of the study, walking ability was found to be significantly lower in LSS individuals compared to healthy individuals.

Santos et al. examined the kinematic and spatiotemporal gait parameters in patients who underwent surgery with a diagnosis of disc herniation or lumbar stenosis before surgery and 1 and 6 months after surgery. As a result of the study, there was an increase in the pelvis, hip and knee range of motion (ROM) after surgery in the disc herniation group, while there was a decrease in the hip ROM values in the stenosis group. It was also observed that the pelvis and hip ROM of both groups remained smaller in the stance phase compared to the control group.

Papadakis et al. examined the changes in gait in patients with lumbar spinal stenosis with the help of an accelerometer before surgery and 6 and 12 months after surgery and showed that there was a significant decrease in the changes in gait in the postoperative period. It was observed that the improvement in the changes in gait was greater in the first month after surgery compared to the 6th and 12th months after surgery.

Purpose of the study:

The study was planned to compare the gait in healthy and patient groups in patients who underwent LSS surgery.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 20-65 and discharged from hospital,
* At least 6 weeks and at most 3 months after surgery,
* No other orthopedic and neurological problems,
* Able to communicate,
* Individuals who agree to participate in the study will be included in the study.

Exclusion Criteria:

* Cognitive impairment,
* Other neurologic, psychiatric and/or orthopedic problems other than lumbar spinal stenosis,
* Medically unstable,
* Individuals with open wounds, circulatory problems, skin lesions in the area to be treated will be excluded from the study.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with spinal stenosis who have undergone surgery
Sampling Method: Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2023-06-13 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of Disability Status (Oswestry Disability Index) | 10 minutes
  It was developed to assess the degree of functional loss in low back pain. The Oswestry Disability Index (OSI), which was shown to be valid and reliable in Turkish in 2004, consists of 10 items. The items question the severity of pain, self-care, lifting and carrying, walking, sitting, standing, sleeping, the degree of change in pain, travel and social life. There are six statements under each item, which the patient marks as appropriate for his/her condition. The first statement is scored as "0", the sixth statement as "5". The score given by the participant to each question is added up. The total score received by the patient is divided by the maximum possible score of 50 points and multiplied by 100 to calculate the percentage. The maximum percentage is "100", the minimum percentage is "0". As the total percentage score increases, the level of disability also increases.
Pain Assessment (Visual Analog Scale-VAS) | 2 minutes
  It is a scale consisting of a single 10 cm line and the pain intensity of patients is evaluated with this scale. Participants are asked to mark the pain intensity at rest and during activity with a pencil on two separate 10 cm lines. The starting point on the scale is expressed as: no pain at all, the last point; the most severe pain encountered in life. When calculating, the distance between the marked point and the starting point is measured in cm with meters. An increase in the score indicates an increase in the intensity of the pain.
Quality of Life Assessment (SF-12) | 5 minutes
  It is a shortened and simplified form of the SF-36 Quality of Life Scale used to assess quality of life. Its Turkish validity and reliability were conducted by Soylu et al. in 2022. The results of the study show that the psychometric properties of the Turkish form of SF-12 are similar to the original version, and therefore it can be used in applications and research to be conducted in our country as an alternative to SF-36. It consists of a total of 12 questions. Each question has its own score. When calculating, 8 sub-items are calculated as percentages, including general health, physical function, physical role difficulty, emotional role difficulty, social function, pain, mental health and vitality. In percentage expressions ranging from 0 to 100, a high percentage indicates good health status.
10 Meter Walk Test | 5 minutes
  It is a test used to evaluate walking. A 10-meter area is determined in advance by the evaluator who will perform the test. The participant is asked to walk at his normal speed along the 10-meter area. When the participant is at the starting line, the stopwatch is started with the start command and the time is stopped when he crosses the finish line. In order to minimize the margin of error, two measurements are taken and the best value is recorded in meters/second (m/s).
BTS G-Walk gait analysis system | 10 minutes
  It is an analysis method that measures all important information such as spatio-temporal parameters of walking, general walking kinematics, spine kinematics and displays this in a computer environment. In the BTS G-Walk walking analysis system, the analysis port is attached to the patient's L5-S1 level and the results are transferred to the computer via the Bluetooth system. With this system; while comparing the walking analysis with normal values in the right and left extremities, it also allows the kinematic analysis of the pelvis to be performed in 3 planes. The resulting reports are created automatically and the system compares directly with the normal range results.

CONTACTS AND LOCATIONS:
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No